CLINICAL TRIAL: NCT00686296
Title: Pilot Study Comparing Taliderm™ Dressing Versus Standard of Care for Open Incision and Drainage of Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-2007-0709-H
Record Dates: First submitted 2008-05-26; First posted 2008-05-29 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Wounds
Keywords: soft tissue abscess requiring incision and drainage
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group II (Active Comparator): Taliderm™ dressing applied until the next scheduled dressing change (up to eight hours), then replaced by a gauze dressing. Gauze dressing changes will continue per standard of care until the scheduled follow-up visits (first or second visit). At the scheduled follow-up visits, the subject will have a Taliderm™ dressing applied and left in place until the next scheduled dressing change (up to eight hours), then will continue standard of care wet to dry gauze dressing changes until next scheduled follow-up visit.
  Interventions: Other: Taliderm™
- III (Other): standard wet to dry dressing with gauze
  Interventions: Other: standard wet to dry dressing with gauze
- group I (Active Comparator): Taliderm™ dressing applied until the next scheduled dressing change (up to eight hours), then replaced by a gauze dressing
  Interventions: Other: Taliderm™

INTERVENTIONS:
Other: Taliderm™ — taliderm™ dressing application once
  Arms: group I
Other: Taliderm™ — Taliderm™ dressing application up to three applications
  Arms: Group II
Other: standard wet to dry dressing with gauze — wet to dry dressing standard of care
  Arms: III

SUMMARY:
To evaluate wound healing with the use of Taliderm™ dressing and compare it to wet to dry dressing in the treatment of open wounds after incision and drainage.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients with soft tissue abscess that will result in an open surgical wounds greater than or equal to 4 cms in any dimension
* Wound will require serial dressing changes
* Greater than or equal to 18 years of age
* Ability to obtain informed consent

Exclusion Criteria:

* Inability to obtain informed consent
* Pregnancy
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study will be rate of wound healing (judged as per cent complete wound closure) at the two (2) and three (3) week follow-up visits. | two and three weeks

SECONDARY OUTCOMES:
occurence of wound infection | two and three weeks

CONTACTS AND LOCATIONS:
Overall Officials: John G Myers, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University Hospital, San Antonio, Texas, United States